CLINICAL TRIAL: NCT04821635
Title: Effects of Training on a Rower Assisted by Electrostimulation of Lower Limbs in Patients With Neurological Disorders (FES-ROW)
Brief Title: Effects of FES-Rowing in Neurological Disorders (FES-ROW)
Acronym: FES-ROW
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participant enrolled
Sponsor: UGECAM Rhône-Alpes (Other)
Collaborators: University of Franche-Comté (Other); Hospices Civils de Lyon (Other); University of Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-1 (FESROW); 2020-A00416-33 (Other: ID-RCB)
Record Dates: First submitted 2021-03-17; First posted 2021-03-29 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-01

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Functional Electrical Stimulation; Cardiovascular Prevention; Neuroplasticity; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rower (Experimental): Single group of 35 traumatic paraplegic patients meeting the inclusion criteria will benefit from the FES-ROW protocol during 9 months
  Interventions: Device: Rower assisted by electrostimulation (FES-ROW)

INTERVENTIONS:
Device: Rower assisted by electrostimulation (FES-ROW) — 1. Pre-inclusion visit
  2. Inclusion visit
  3. Phase 1 Rower-FES with lower limbs (Month 0 to Month 3: M0-M3):
     Training on a rower with solicitation of the electrostimulated lower limbs only for a period of 3 months at the rate of 3 sessions of 30 minutes per week
  4. Interim assessment visit at Month 3 (M3)
  5. Phase 2 Rower-FES with lower limbs + upper limbs (Month 3 to Month 6: M0-M6):
     Training on with solicitation of the electrostimulated lower and upper limbs for a period of 3 months at the rate of 3 sessions of 30 minutes per week
  6. Final assessment visit at Month 6 (M6)
  7. End of clinical research visit, 3 months after the end of training (Month 9, M9)

SUMMARY:
The main objective of this project is to measure the increase in aerobic physical and metabolic capacities with a 6-month training on a rower assisted by electrostimulation of lower limbs in a population of adults with traumatic paraplegia.

DETAILED DESCRIPTION:
Beyond the inability to walk, chronic paraplegic patients show an increase in their mortality from cardiovascular pathologies, compared to the same age groups of the general population. It is the hypoactivity induced by neurological impairment that is implicated in the first place in the pathogenesis of these abnormalities. The search for training methods adapted to these patients is justified to limit cardiovascular morbidity and mortality.

The aim of this project is to measure the increase in aerobic physical and metabolic capacities with a 6-month training on a rower assisted by electrostimulation of lower limbs in a population of adults with stabilized paraplegia (non-walkers), of traumatic origin.

Study is divided in two 3-month phases. The first consists on a training on a rowing machine with solicitation of the electrostimulated lower limbs only for a period of 3 months at the rate of 3 sessions of 30 minutes per week. The second consists on a training on a rowing machine with solicitation of the electrostimulated lower limbs and upper for a period of 3 months at the rate of 3 sessions of 30 minutes per week. The evaluations are composed of the measurement of maximum oxygen consumption, muscle and neurological parameters

ELIGIBILITY:
Inclusion Criteria:

* Paraplegia with traumatic origin
* Spinal cord injury AIS (ASIA Impairment Scale) score A and B at least 12 months old
* Patient having given written consent
* Patient with social security scheme
* Ability to obtain a leg extension with a 30-minute electrostimulation program

Exclusion Criteria:

* Protected adults (person in guardianship, curators or legal protection)
* Presence of contraindication criteria to carrying out a stress test or sustained physical activity decided by the doctor following the person with spinal cord injury.
* Drug treatment with cardiovascular or antidepressant effect
* Pressure sore
* Other associated neurological pathologies (stroke, peripheral neuropathy, myopathy, head trauma, ...)
* Affection of the shoulders of any etiology that could compromise the ability to use the rower.
* Spasticity of the lower limbs: Modified Ashworth Scale (MAS) greater than or equal to 2/4 (specifically quadriceps / Hamstrings)
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
VO2 peak at 6 months (L/min) | 6 months
  Comparison of the maximum oxygen consumption (VO2 peak in L/min) measured during an incremental maximum stress test on a hand ergometer between the end of training on a rower (M6) and inclusion (M0).

SECONDARY OUTCOMES:
VO2 peak at 3 and 9 months (L/min) | 9 months
  Comparison of the maximum oxygen consumption (VO2 peak in L/min) measured during an incremental maximum stress test on a hand ergometer between the end of first training phase (M3) and inclusion (M0) and between the end of the study (M9) and inclusion (M0).
First ventilatory threshold in the VO2max test at 0, 3, 6 and 9 months (L/min) | 9 months
  Comparison of the first ventilatory threshold (in L/min) in the VO2max test measured during an incremental maximum stress test on a hand ergometer between the end of first training phase (M3), the end of second phase (M6), the end of the study (M9) and inclusion (M0).
Maximum electro-induced force at 0, 3, 6 and 9 months (Nm) | 9 months
  Comparison of maximum electro-induced force (in Newton) assessment with a device for measuring the force of the knee extensor muscles between the end of first training phase (M3), the end of second phase (M6), the end of the study (M9) and inclusion (M0).
Thigh perimeter at 0, 3, 6 and 9 months (cm) | 9 months
  Comparison of thigh perimeter (in cm) assessment between the end of first training phase (M3), the end of second phase (M6), the end of the study (M9) and inclusion (M0).
Maximum power at 0, 3, 6 and 9 months (Watts) | 9 months
  Comparison of the maximum power (in Watts) developed during the stress test on a hand ergometer between the end of first training phase (M3), the end of second phase (M6), the end of the study (M9) and inclusion (M0).
Response to stimulation at 0, 3, 6 and 9 months (mA) | 9 months
  Comparison of the minimum threshold (Intensity in mA) of response to stimulation of the extensor muscles of the knee between the end of first training phase (M3), the end of second phase (M6), the end of the study (M9) and inclusion (M0).
Assessment of spasticity at 0, 3, 6 and 9 months | 9 months
  Assessment of spasticity with Ashworth scale (rating from 0 to 4 which is the worst score) and Pendulum test (rating from 1 to 5 which is the worst score) between the end of first training phase (M3), the end of second phase (M6), the end of the study (M9) and inclusion (M0).
Intensity of osteotendinous reflexes at 0, 3, 6 and 9 months | 9 months
  Comparison of the intensity of osteotendinous reflexes (Absent, normal and lively / diffuse / polykinetic) between the end of first training phase (M3), the end of second phase (M6), the end of the study (M9) and inclusion (M0).
Self-assessment at 0, 3, 6 and 9 months | 9 months
  Self-assessment with Goal Attainment Scaling (GAS) between the end of first training phase (M3), the end of second phase (M6), the end of the study (M9) and inclusion (M0).
  GAS rating is divided in 5 levels:
  * -2: Current level
  * -1: Improvement
  * 0: Expected level after action
  * +1: Level better than expected
  * +2: Maximum level expected
ASIA (American Spinal Injury Association) score at 0, 6 and 9 months | 9 months
  Comparison between the end of the study following the remanence period (M9) and the inclusion (M0) and M6 of the parameters of ASIA (American Spinal Injury Association) score.

CONTACTS AND LOCATIONS:
Overall Officials: Julie R Di Marco, M.D, Principal Investigator — UGECAM SSR Val Rosay
Locations (2):
- France (2):
  - HIA Desgenettes, Lyon, Rhône
  - SSR Val Rosay UGECAM, Saint-Didier-au-Mont-d'Or, Rhône

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheeler GD, Andrews B, Lederer R, Davoodi R, Natho K, Weiss C, Jeon J, Bhambhani Y, Steadward RD. Functional electric stimulation-assisted rowing: Increasing cardiovascular fitness through functional electric stimulation rowing training in persons with spinal cord injury. Arch Phys Med Rehabil. 2002 Aug;83(8):1093-9. doi: 10.1053/apmr.2002.33656. PMID 12161830
- [Background] Popovic-Maneski L, Aleksic A, Metani A, Bergeron V, Cobeljic R, Popovic DB. Assessment of Spasticity by a Pendulum Test in SCI Patients Who Exercise FES Cycling or Receive Only Conventional Therapy. IEEE Trans Neural Syst Rehabil Eng. 2018 Jan;26(1):181-187. doi: 10.1109/TNSRE.2017.2771466. PMID 29324409
- [Background] Deley G, Denuziller J, Babault N. Functional electrical stimulation: cardiorespiratory adaptations and applications for training in paraplegia. Sports Med. 2015 Jan;45(1):71-82. doi: 10.1007/s40279-014-0250-2. PMID 25205000